CLINICAL TRIAL: NCT01894100
Title: Defining and Correcting Limb Length Inequality in Adults With Knee or Hip Symptoms
Brief Title: Shoe Lifts for Leg Length Inequality in Adults With Knee or Hip Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Yvonne Golightly PT, PhD, Research Assistant Professor, Epidemiology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0807
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Leg Length Inequality; Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Leg Length Inequality; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Intervention Group (Other): This group will not receive shoe lifts during the first 3 months after baseline. At 3 months, they will begin the shoe lift correction for leg length inequality.
  Interventions: Device: Shoe lift correction for leg length inequality
- Immediate Intervention Group (Experimental): At baseline, participants in this group will begin shoe lift correction for leg length inequality.
  Interventions: Device: Shoe lift correction for leg length inequality

INTERVENTIONS:
Device: Shoe lift correction for leg length inequality — Lift therapy will be administered by a physical therapist. Heel lifts and full length inserts used inside participants' shoes will be constructed on-site. If an external shoe lift is required for a participant, a local shoe repair shop will construct the lifts and add them to the outside of the shoe. Participants will be required to wear the lift in their shoes when they are walking or standing while enrolled in the study; participants will keep a daily diary to record their compliance (number of hours lift worn per day, amount of lift used, type of shoes worn, general symptoms experienced, and activities performed). They will be contacted weekly to be reminded to increase their lift height and identify when they have achieved their optimal lift height.

SUMMARY:
Limb length inequality is when a person has one leg that is longer than the other. This research will look at correcting limb length inequality in adults with knee or hip symptoms. This study will examine whether ways of measuring leg length inequality in the clinic are valid and reliable, determine whether foot posture (flat foot, normal, and high arch) is related to leg length inequality, and determine whether shoe lifts are a helpful treatment for leg length inequality and knee/hip symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to examine the optimal clinical assessment method(s) for leg length inequality (LLI), determine if there is an association between foot posture (flat foot, normal, and high arch) and LLI, and gather preliminary data on lift therapy as a treatment for LLI and knee/hip symptoms. The specific aims of the project are as follows:

Specific Aim 1: Determine the validity and reliability of 4 clinical methods for assessing LLI.

Specific Aim 2: Determine differences in static and dynamic foot postures between longer and shorter limbs.

Specific Aim 3: Assess the feasibility of conducting a specific lift therapy intervention among individuals with a LLI and knee or hip pain, refining procedures as needed.

Public Health Impact: Results from the proposed research will be used to: 1) improve diagnosis of LLI by providing evidence on the various assessment methods for the clinicians who most frequently use clinical methods (i.e., physical therapists, chiropractors, podiatrists, and primary care physicians), and 2) develop and test new non-pharmacologic/non-invasive intervention strategies aimed at reducing pain and improving function in individuals with osteoarthritis and LLI.

ELIGIBILITY:
Inclusion Criteria:

* participants from the Johnston County Osteoarthritis Project who have been previously identified to have a LLI and knee or hip symptoms

Exclusion Criteria:

* hospitalized for stroke, myocardial infarction, coronary artery revascularization, or diagnosis of metastatic cancer in the past 3 months
* terminal illness
* rheumatoid arthritis, severe fibromyalgia, or other systemic rheumatic disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M Golightly, PT, MS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-CH Thurston Arthritis Research Center, Smithfield, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning 6/14/2013, 510 participants from the Johnston County Osteoarthritis Project cohort were identified as potential participants for this study based on a history of knee or hip symptoms and a body mass index of <35 kg/m2 at last cohort study visit.
Pre-assignment Details: Of the 510 participants that research assistants attempted to contact via telephone, 46 participants were eligible and agreed to participate in the study (enrolled from 8/7/2013 through 4/30/2014). 16 were excluded from assignment to an intervention group because they did not have a leg length inequality >=1/8 inch on standing radiograph.
Period: Overall Study
Arm/Group | Delayed Intervention Group | Immediate Intervention Group
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Intervention Group | Immediate Intervention Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8) | 70 (8) | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score [Mean (Standard Deviation); unit: units on a scale] — Possible scores range from 0-96 (no problems to extreme problems)
  units on a scale | 34.8 (11.4) | 37.7 (11.1) | 36.2 (8.4)
WOMAC Pain [Mean (Standard Deviation); unit: units on a scale] — Possible scores range from 0-20 (no pain to extreme pain)
  units on a scale | 8.0 (2.5) | 8.7 (2.5) | 8.4 (2.5)
WOMAC Stiffness [Mean (Standard Deviation); unit: units on a scale] — Possible score range from 0-8 (no stiffness to extreme stiffness)
  units on a scale | 3.1 (1.6) | 3.8 (0.8) | 3.4 (1.3)
WOMAC Function [Mean (Standard Deviation); unit: units on a scale] — Possible scores range from 0-68 (no problems to extreme problems with function).
  units on a scale | 23.7 (9.1) | 25.1 (9.0) | 24.4 (8.9)
8 foot walk [Mean (Standard Deviation); unit: seconds] | 3.5 (0.9) | 3.8 (1.1) | 3.7 (1.0)
5 timed chair stands [Mean (Standard Deviation); unit: seconds] | 18.9 (11.0) | 18.4 (8.5) | 18.7 (9.6)
single leg stance [Mean (Standard Deviation); unit: seconds] | 6.8 (3.7) | 5.4 (4.0) | 6.1 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Western Ontario and McMasters Universities Osteoarthritis Index pain subscale is a 5 item questionnaire that asks participants to rate their pain during walking, using stairs, in bed, sitting or lying, and standing. Each item is rated by the participant as 0-4 (no pain to extreme pain). Total scores on the pain subscale range from 0 to 20 (no pain to extreme pain).
Time Frame: Baseline and 3 months after initiating intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Delayed Intervention Group | Immediate Intervention Group
Number analyzed (Participants) | 13 | 15
units on a scale | -0.8 (3.6) | -2.9 (3.4)

2. Secondary Outcome: Change in Lower Extremity Physical Function
Description: For self-reported lower extremity physical function: Western Ontario and McMasters Universities Osteoarthritis Index physical function subscale. The physical function subscale includes 17 items that ask about difficulty with stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, and light household duties. Participants rate each item on a scale of 0-4 (no difficulty to extreme difficulty. Totals scores for this subscale range from 0-68 (no difficulty to extreme difficulty).
Time Frame: Baseline and 3 months post intervention
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Delayed Intervention Group | Immediate Intervention Group
Number analyzed (Participants) | 15 | 15
units on scale | -2.9 (6.9) | -9.5 (6.5)

ADVERSE EVENTS:
Time Frame: Full study period for both groups: 6 months for Delayed Intervention Group and 9 months for Immediate Intervention Group
Arm/Group | Delayed Intervention Group | Immediate Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Intervention Group (N=15) | Immediate Intervention Group (N=15)
redness of skin of big toe (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant with redness of skin on big toe from pressure inside toe case of shoe with full length shoe lift. Symptom was relieved when full length shoe lift was changed to heel lift, allowing more space for the big toe in the toe case of the shoe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No